CLINICAL TRIAL: NCT02599948
Title: FRench-speAking Icu (Intensive Care Unit) Nutritional Survey
Acronym: FRANS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00003835
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2014-08

CONDITIONS: Intensive Care Units (ICUs)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients hospitalised in ICU: Patients hospitalised in ICU
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Assessment of nutritional practices in french intensive care units.

DETAILED DESCRIPTION:
Assessment of nutritional practices in french intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized patients in intensive care units for an expected period of stay> 3 days

Exclusion Criteria:

* Refuse to participate in the Protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized patients in ICU
Sampling Method: Non-Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Frequency of patients receiving parenteral nutrition within the first 10 days after ICU admission | 10 days

REFERENCES:
- [Result] Pardo E, Lescot T, Preiser JC, Massanet P, Pons A, Jaber S, Fraipont V, Levesque E, Ichai C, Petit L, Tamion F, Taverny G, Boizeau P, Alberti C, Constantin JM, Bonnet MP; FRANS study group. Association between early nutrition support and 28-day mortality in critically ill patients: the FRANS prospective nutrition cohort study. Crit Care. 2023 Jan 7;27(1):7. doi: 10.1186/s13054-022-04298-1. PMID 36611211